CLINICAL TRIAL: NCT02869204
Title: The Effect of L-PRP on Wound Healing and Wound Infection After Pancreaticoduodenectomy / Whipples Surgery
Brief Title: The Effect of a Local Injection of a Platelet Concentrate on Infection and Healing of Surgical Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, MD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-16025526
Record Dates: First submitted 2016-08-03; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Wound Infection and Wound Healing
MeSH Terms: conditions — Wound Infection | interventions — Ascorbic Acid; Zinc; Arginine

ARMS (2):
- Leucocyte - Platelet rich Plasma and Dietary Supplements (Experimental): An application of an autologous platelet concentrate (20 ml). This is injected once, locally in the muscle after closure of the inner fascia and before closure of the outer fascia.
  A daily dietary supplement of Vitamin C, Zinc and L-Arginine. Provided from POD2-3 until POD30
  Interventions: Other: Leucocyte - Platelet rich Plasma; Dietary Supplement: Vitamin C; Dietary Supplement: Zinc; Dietary Supplement: L-Arginine
- Treatment as usual (No Intervention): Patients are treated as usual.

INTERVENTIONS:
Other: Leucocyte - Platelet rich Plasma — Autologous L-PRP are studied regarding it's accelerating effect on tissue repair.
  Other Names: L-PRP
  Arms: Leucocyte - Platelet rich Plasma and Dietary Supplements
Dietary Supplement: Vitamin C — A daily dietary supplement of 500 mg Vitamin C. Provided from POD2-3 until POD30
  Arms: Leucocyte - Platelet rich Plasma and Dietary Supplements
Dietary Supplement: Zinc — A daily dietary supplement of 44 mg Zinc. Provided from POD2-3 until POD30
  Arms: Leucocyte - Platelet rich Plasma and Dietary Supplements
Dietary Supplement: L-Arginine — A daily dietary supplement of 5 g L-Arginine. Provided from POD2-3 until POD30
  Arms: Leucocyte - Platelet rich Plasma and Dietary Supplements

SUMMARY:
The purpose of this project is to investigate whether a combination of a local injection of platelet rich plasma (PRP) combined with a daily supplement of vitamin C, zinc, L-arginine, as well as high protein diet (1.5 g of protein per kilo body weight per day) can promote tissue healing in patients undergoing open upper-abdominal surgery.

Primary endpoint is cases of wound infection and secondary endpoints are time of tissue regeneration (days), judged by traditional clinical observation and experimentally assessed by ultrasound.

The experiment is performed as a parallel two-armed, randomized, controlled trial.

A total of 40 subjects will be included in the trial i order to ensure the power of the study, despite a drop off of up to 25%.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Rigshospitalets Surgical gastroenterology clinic
* Planned to have a Pancreaticoduodenectomy preformed
* Being able to understand Danish, the trial and what it means to be enrolled in the trial
* Capable of signing a written consent
* Living i the Regional Capital (excl. Bornholm) or the Regional of Sjælland (north of Næstved)

Exclusion Criteria:

* Dysregulated diabetes mellitus type I or II
* Alcohol consumption above 14 or 7 x 12 g alcohol per week (men vs women)
* Participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with wound infection assessed by traditional clinical observation of the cicatrice | From date of surgery until the date of first documented event of infection or date of death from any cause, whichever came first, assessed up to 30 days .
  Infection are defined as a collection of pus in the wound that require revision.
  It is assessed by observation from the hospital staff.

SECONDARY OUTCOMES:
Number of days before the surgical wound are full epithelized assessed by observation of the cicatrice | Up to 30 days
  Digital photos of the cicatrice will be collected and analyzed for the amount of remaining scab.
Other postoperative complications | Up to 30 days
Length of stay (LOS) | 30 days
Experience of pain assessed by a VAS (Visual analogue scale) | Up to 30 days
Mobilization assessed by "Timed Up & Go (TUG)" | Up to 30 days
  Timed Up & Go, also known as TUG, measures the time it takes a study subject to stand up, walk 3 meters, turn around, walk back and sit down.
Inflammatory responds assessed by blood sample analysis of the acute phase reactant CRP (c-reactive protein) | Up to 30 days
Inflammatory responds assessed by blood sample analysis of the acute phase reactant leucucytes | Up to 30 days